CLINICAL TRIAL: NCT02536170
Title: Phase 2 Randomized Control Trial of Arginine Therapy for Pediatric Sickle Cell Disease Pain
Brief Title: Arginine Therapy for Sickle Cell Disease Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Claudia R. Morris, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00076988; FD-R-004814 (Other Grant/Funding Number: FDA); 1K24AT009893-01 (NIH)
Record Dates: First submitted 2015-08-27; First posted 2015-08-31 (Estimated); Results first posted 2022-06-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Pain Episode
Keywords: Arginine Therapy
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- L-Arginine (Experimental): Participants will be randomized to receive an intravenous (IV) infusion of L-arginine (100 mg/kg) three times a day until time of discharge from the emergency department (ED) or hospital.
  Interventions: Drug: L-arginine
- Loading Dose and L-Arginine (Experimental): Participants will be randomized to receive an intravenous (IV) infusion of one-time loading dose of L-arginine (200 mg/kg) followed by standard dose (100 mg/kg) three times a day until time of discharge from the emergency department (ED) or hospital.
  Interventions: Drug: L-arginine; Drug: L-arginine Loading Dose
- Placebo (Placebo Comparator): Participants will be randomized to receive an intravenous (IV) infusion of placebo (normal saline 1-2 ml/kg) three times a day until time of discharge from the emergency department (ED) or hospital.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L-arginine — L-arginine will be dispensed intravenously (IV) in the standard dose of 100 mg/kg three times a day until discharge from the emergency department (ED) or hospital.
  Other Names: Arginine
  Arms: L-Arginine; Loading Dose and L-Arginine
Drug: L-arginine Loading Dose — One loading dose of L-arginine will be dispensed intravenously (IV) at 200 mg/kg
  Other Names: Arginine
  Arms: Loading Dose and L-Arginine
Other: Placebo — Placebo of intravenous (IV) normal saline 1-2 ml/kg three times a day until discharge from the emergency department (ED) or hospital.
  Arms: Placebo

SUMMARY:
The aim of this study is to determine whether giving extra arginine, a simple amino acid, to patients with sickle cell disease seeking treatment for a pain crisis (vaso-occlusive painful events (VOE) will decrease pain scores, decrease the need for pain medications or decrease length of hospital stay or emergency department visit. Funding Source - FDA OOPD.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of IV L-arginine hydrochloride therapy in children with sickle cell disease (SCD) and vaso-occlusive pain events (VOE). Specifically, the impact on total opioid use (mg/kg) over the duration of their emergency department (ED) visit and hospital stay will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of sickle cell disease (SCD); all genotypes
* Pain requiring medical care in an acute care setting (such as the emergency department or ED, hospital ward, day hospital, clinic) not attributable to non-sickle cell causes, that is moderate-to-severe requiring parenteral opioids

Exclusion Criteria:

* Decision to discharge home from the acute care setting
* Hemoglobin less than 5 gm/dL or immediate need for red cell transfusion anticipated within next 12 hours
* Hepatic dysfunction of SGPT greater than 3 times the upper value
* Renal dysfunction of creatinine greater than 1.0
* Mental status or neurological changes
* Acute stroke or clinical concern for stroke
* Pregnancy
* Allergy to arginine
* Two (2) or more ED visits for VOE within the last 7 days prior to CURRENT ED visit
* Hospitalization within 14 days
* Previous randomization in this arginine RCT (patient consented and screen failed before receiving study drug or placebo remains eligible for future participation).
* Use of inhaled nitric oxide, sildenafil or arginine within the last month
* PICU admission from the emergency department
* Hypotension requiring treatment with clinical intervention
* Acidosis with Co2≤ 16
* Newly started on HU for <3 months
* Not an appropriate candidate in the investigator's judgment
* Patient refusal

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2016-02; Primary Completion 2021-02-21 (Actual); Study Completion 2021-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Morris, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Children's Healthcare of Atlanta at Hugh Spalding, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakshi N, Liu Z, Gillespie S, Keesari R, Leake D, Khemani K, Kumari P, Rees CA, Dampier C, Morris CR. Patient-reported outcomes in children with sickle cell disease at presentation for an acute pain episode. Blood Adv. 2023 Sep 12;7(17):5103-5107. doi: 10.1182/bloodadvances.2021006794. No abstract available. PMID 36322873
- [Result] Reyes LZ, Figueroa J, Leake D, Khemani K, Kumari P, Bakshi N, Lane PA, Dampier C, Morris CR. Safety of intravenous arginine therapy in children with sickle cell disease hospitalized for vaso-occlusive pain: A randomized placebo-controlled trial in progress. Am J Hematol. 2022 Jan 1;97(1):E21-E24. doi: 10.1002/ajh.26396. Epub 2021 Nov 12. No abstract available. PMID 34724240
- [Derived] Morris CR, Hatabah D, Korman R, Gillespie S, Bakshi N, Brown LA, Harris F, Leake D, Rees CA, Khemani K, Vichinsky EP, Locke A, Wynn B, Griffiths MA, Wilkinson H, Kumari P, Sudmeier L, Shiva S, Dampier CD. Arginine Therapy for Pain in Sickle Cell Disease: A Phase-2 Randomized, Placebo-Controlled Trial. Am J Hematol. 2025 Jul;100(7):1119-1131. doi: 10.1002/ajh.27692. Epub 2025 Apr 24. PMID 40270092
- [Derived] Morris CR, Brown LAS, Reynolds M, Dampier CD, Lane PA, Watt A, Kumari P, Harris F, Manoranjithan S, Mendis RD, Figueroa J, Shiva S. Impact of arginine therapy on mitochondrial function in children with sickle cell disease during vaso-occlusive pain. Blood. 2020 Sep 17;136(12):1402-1406. doi: 10.1182/blood.2019003672. PMID 32384147

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Started | 36 | 36 | 36
Completed | 36 | 36 | 36
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo | Total
Number analyzed (Participants) | 36 | 36 | 36 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 31 | 35 | 100
  Between 18 and 65 years | 2 | 5 | 1 | 8
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.49 (3.76) | 13.63 (3.7) | 12.27 (4.0) | 13.13 (3.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 20 | 56
  Male | 17 | 19 | 16 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 36 | 36 | 35 | 107
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 36 | 36 | 36 | 108
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 36 | 108

OUTCOME MEASURES:

1. Primary Outcome: Total Parenteral Opioid Use in IV Morphine Equivalents
Description: The total amount of parenteral opioids used by participants measured in mg/kg of IV morphine equivalents. The total is calculated after study drug delivery for participants in the emergency department (ED) and during hospital stay.
Time Frame: Post study drug delivery to discharge from the hospital (Up to 8 days)
Measure: Mean (Standard Deviation); unit: mg/Kg
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
mg/Kg | 1.77 (1.91) | 1.95 (2.09) | 2.36 (3.14)

2. Secondary Outcome: Length of Hospital Stay
Description: The total number of hours spent in the hospital from study drug delivery to time of discharge.
Time Frame: Discharge (Up to 8 days)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
hours | 71.3 (50.8) | 76.9 (49.9) | 84.9 (90.5)

3. Secondary Outcome: Time to Vaso-occlusive Pain Event (VOE) Resolution in Emergency Department
Description: The total number of hours between study drug delivery and the last parenteral opioid.
Time Frame: Post study drug delivery (Up to 8 hours)
Population: Time to vaso-occlusive pain event (VOE) resolution in emergency department could not be determined as none of the participants had pain resolution in the Emergency department and were hospitalized
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
hours | NA (NA) — Time to vaso-occlusive pain event (VOE) resolution in emergency department could not be determined as none of the participants had pain resolution in the Emergency department and were hospitalized | NA (NA) — Time to vaso-occlusive pain event (VOE) resolution in emergency department could not be determined as none of the participants had pain resolution in the Emergency department and were hospitalized | NA (NA) — Time to vaso-occlusive pain event (VOE) resolution in emergency department could not be determined as none of the participants had pain resolution in the Emergency department and were hospitalized

4. Secondary Outcome: Time to Vaso-occlusive Pain Event (VOE) Resolution in Hospital
Description: The total number of hours between study drug delivery and time of last parenteral opioid use, pain relief improved to tolerate oral pain medications
Time Frame: Post study drug delivery until discharge (up to 8 days)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
hours | 57.3 (50.8) | 55.1 (42.9) | 69.3 (85.1)

5. Secondary Outcome: Change in Vaso-occlusive Pain (VOE) Scores
Description: Pain associated with VOE will be measured on a scale of 0-10, by asking subjects to rate their pain level on a subjective scale from 0 to 10, with the ends representing the extreme limits of "no-pain" (0) and "worst pain" (10).
Time Frame: Baseline, Time of discharge (Up to 8 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
score on a scale
  Emergency Department (ED) arrival Pain Score | 8.89 (1.01) | 8.86 (1.46) | 8.86 (1.36)
  Time of hospital discharge Pain Score | 4.5 (3.46) | 4.75 (3.35) | 4.56 (2.97)
  Hospital Discharge Minus ED Arrival | -4.39 (3.41) | -4.11 (3.54) | -4.31 (3.09)

6. Secondary Outcome: Length of Emergency Department (ED) Stay
Description: Total hours from time of ED triage to ED discharge or hospital admission.
Time Frame: Until discharge or Hospital Admission (Up to 24 hours)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
hours | 6.29 (15.84) | 5.67 (12.33) | 4.08 (4.26)

7. Secondary Outcome: Rate of Emergency Department (ED) Discharge
Description: Number of participants discharged from ED without a hospital ward admission.
Time Frame: Post emergency department admission (Up to 24 hours)
Population: All patients were admitted to the hospital, none was discharged during Emergency Department stay.
Measure: Count of Participants; unit: Participants
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
Participants | 0 | 0 | 0

8. Secondary Outcome: Total Opioid Dose (ORAL + Parenteral) in mg/kg IV Morphine Equivalents
Description: Total opioid dose (ORAL + Parenteral) in mg/kg IV morphine equivalents after study drug delivery up to hospital discharge (up to 8 days)
Time Frame: Post study drug delivery up to hospital discharge (Up to 8 days)
Measure: Mean (Standard Deviation); unit: mg/Kg
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
mg/Kg | 2.11 (2.18) | 2.35 (2.19) | 2.82 (3.65)

9. Secondary Outcome: Total Number of Study Drug Doses
Description: The total number of study drug doses given throughout the study period.
Time Frame: Duration of study (Up to 8 days)
Measure: Number; unit: doses
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
doses | 298 | 330 | 329

10. Secondary Outcome: Rate of Acute Chest Syndrome
Description: Number of participants who develop acute chest syndrome (not diagnosed prior to study drug delivery) throughout the study period.
Time Frame: Duration of study (Up to 8 days)
Measure: Count of Participants; unit: Participants
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
Participants | 4 | 3 | 1

11. Secondary Outcome: Rate of Blood Transfusion
Description: Number of participants requiring a blood transfusion throughout the study period.
Time Frame: Duration of study (Up to 8 days)
Measure: Count of Participants; unit: Participants
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
Participants | 3 | 2 | 5

12. Secondary Outcome: Oxygen Saturation Level
Description: Average oxygen saturation level of participants at time of ED arrival
Time Frame: At time of Emergency Department Admission
Measure: Mean (Standard Deviation); unit: percentage of oxygenated hemoglobin
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
percentage of oxygenated hemoglobin | 95.5 (14.8) | 98 (1.96) | 98.1 (2.14)

13. Secondary Outcome: Oxygen Saturation Level
Description: The difference in oxygen saturation levels from emergency department arrival to hospital discharge.
Time Frame: At time of hospital admission and at time of Hospital discharge (Up to 8 days)
Measure: Mean (Standard Deviation); unit: percentage of oxygenated hemoglobin
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
percentage of oxygenated hemoglobin
  Oxygen saturation measures at time of emergency Department arrival | 95.5 (14.8) | 98 (1.96) | 98.1 (2.14)
  Oxygen saturation at Hospital Discharge | 98 (2.75) | 98.6 (2.11) | 98.4 (2.02)

14. Secondary Outcome: Rate of Return Visits to Emergency Department (ED) Within 72 Hours
Description: Number of ED visits from patients who have been discharged within the previous 72 hours.
Time Frame: Post hospital discharge (within 72 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
Participants | 0 | 0 | 0

15. Secondary Outcome: Rate of Hospital Re-admissions Within 72 Hours
Description: Number of patients readmitted to the hospital within 72 hours of discharge.
Time Frame: Post hospital discharge (within 72 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
Participants | 2 | 2 | 2

16. Secondary Outcome: Rate of Return Visits to Emergency Department (ED) Within 30 Days
Description: Number of ED visits from patients who have been discharged within the previous 30 days.
Time Frame: Post hospital discharge (within 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
Participants | 0 | 1 | 0

17. Secondary Outcome: Rate of Hospital Re-admissions With 30 Days
Description: Number of patients readmitted to the hospital within 30 days of discharge.
Time Frame: Post hospital discharge (within 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
Number analyzed (Participants) | 36 | 36 | 36
Participants | 2 | 7 | 4

ADVERSE EVENTS:
Time Frame: Information on adverse events will be assessed from the time study participation begins through the end of study follow up (up to 30 days, or after 21 doses or until discharge, whichever comes first).
Arm/Group | L-Arginine | Loading Dose and L-Arginine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 4/36 | 9/36 | 6/36
Other Adverse Events (participants affected / at risk) | 30/36 | 31/36 | 30/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-Arginine (N=36) | Loading Dose and L-Arginine (N=36) | Placebo (N=36)
Re-admission: Acute Chest Syndrome (Cardiac disorders) | 1 (1) | 2 (2) | 1 (2)
Re-admission: Vaso-Occlusive Pain Event (Vascular disorders) | 2 (3) | 7 (13) | 3 (4)
Re-admission: Non sickle Cell event (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Prolonged hospitalization: Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Prolonged hospitalization: Priapism (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-Arginine (N=36) | Loading Dose and L-Arginine (N=36) | Placebo (N=36)
Acute Chest Syndrome after randomization (Cardiac disorders) | 4 (4) | 3 (3) | 1 (1)
Acute Chest Syndrome (Cardiac disorders) | 4 (4) | 4 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6) | 10 (10)
Oxygen administered (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (5)
Headache (Nervous system disorders) | 14 (16) | 10 (10) | 9 (9)
Headache after randomization (Nervous system disorders) | 7 (7) | 4 (4) | 5 (5)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 6 (6) | 5 (5) | 5 (5)
Fever (General disorders) | 7 (7) | 10 (10) | 6 (6)
Anorexia (Gastrointestinal disorders) | 10 (10) | 8 (8) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 9 (9) | 9 (9) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 15 (15) | 17 (17) | 13 (13)
Vomiting (Gastrointestinal disorders) | 9 (9) | 11 (12) | 8 (8)
Vomiting after randomization (Gastrointestinal disorders) | 8 (8) | 5 (5) | 5 (5)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Leg/ Neck/ Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Splenic Sequestration (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lip Swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Transfusion (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 5 (5)
Emergency Department visit after Discharge (General disorders) | 0 (0) | 1 (2) | 0 (0)
Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Elevated ALT (Blood and lymphatic system disorders) | 5 (5) | 5 (5) | 4 (4)
Elevated AST (Blood and lymphatic system disorders) | 6 (6) | 9 (9) | 7 (7)
Elevated Bilirrubin (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 2 (2)
Elevated Alkaline Phosphatase (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Elevated creatinine (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0)
Decreased Neutrophil count (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia/ Decreased Hemoglobin (Blood and lymphatic system disorders) | 7 (7) | 7 (7) | 8 (8)
Hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Decreased Platelet count (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased Bicarbonate (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/70/NCT02536170/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT02536170/ICF_001.pdf